CLINICAL TRIAL: NCT05501093
Title: Diabetes Reversal and the Subgingival Microbiota
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Temple University (Other); Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 825975; 1R01DE026603-01A1 (NIH)
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Diabetes type2; Bariatric Surgery Candidate
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Oral plaque was collected with the use of a microbrush, small paper points and periopaper strips.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic patients: Diabetic patients who plan to undergo bariatric surgery
  Interventions: Other: sample collection
- Normo-glycemic (non-diabetic) patients: Non-diabetic patients who plan to undergo bariatric surgery
  Interventions: Other: sample collection

INTERVENTIONS:
Other: sample collection — Blood, plaque, and other oral samples

SUMMARY:
This study seeks to examine the impact of bariatric surgery on oral bacteria in diabetic compared to non-diabetic patients. The purpose of this research study is to examine how diabetes changes the bacteria in the mouth. This is an important question since bacterial changes may impact oral health. Participants will attend a screening and baseline visit prior to bariatric surgery and three post bariatric surgery appointments (3 weeks post, 6 months post and 1 year to 18 months post). Samples collected at each study visit include blood, plaque, and other oral samples. At the last study visit there is an optional dental cleaning.

ELIGIBILITY:
Inclusion Criteria:

* Men and women undergoing bariatric surgery who are 25-65 years old.
* BMI > 35 kg/m2.
* Diabetic subjects: HbA1c> 6.0% or fasting plasma glucose >126 mg/dl).
* Normoglycemic subjects: HbA1c<5.75% or fasting plasma glucose <100 mg/dl).
* Dental criteria: Minimum of 4 posterior teeth.
* Signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Subjects diagnosed with type 1 diabetes, maturity onset diabetes of the young (MODY), or latent autoimmune diabetes in adults (LADA).
* Women who are considering pregnancy or are currently breastfeeding.
* Individuals with a history of chronic inflammatory or autoimmune diseases or taking medications that affect immune function or affect body weight such as chronic systemic steroids.
* Currently smoke more than 10 cigarettes per day.
* Periodontal treatment within 3 months of bacterial sampling.
* Acute periodontal infection (abscess) within 1 month of bacterial sampling or abscess in teeth or adjacent teeth within 1 month of sampling.
* Treatment with antibiotics within one month of sample collection (except as part of the surgical regimen of prophylactic antibiotic immediately prior to surgery).
* A treatment regimen of steroids within 1 month of sample collection.

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study participants will be men and women, 25-65 years old, with a Body Mass Index (BMI) of ≥35 kg/m2 who are scheduled to undergo bariatric surgery at the University of Pennsylvania or Temple University for treatment of obesity or obesity and type 2 diabetes. The total target enrollment is 130 diabetic and 104 normoglycemic subjects.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Bacterial composition | 18 months
  as determined by 16s rRNA community profiling

SECONDARY OUTCOMES:
Bacterial mRNA profiling | 18 months
  RNA will be isolated then amplified by the MessageAmp II bacterial RNA amplification kit (Ambion/Life Technologies). Ribosomal RNA will be depleted with the RiboZero human/mouse and meta bacterial kits (Epicentre/Illumina) and human mRNA will be depleted with oligo(dT). Illumina sequencing libraries will be constructed with the Illumina TruSeq RNA kit and assessed with an Illumina HiSeq instrument.
Gingival inflammation | 18 mos.
  samples will be assessed for inflammatory cytokines (e.g. IL-1β, IL-17 or TNF) by multiplex assay or ELISA assay

CONTACTS AND LOCATIONS:
Overall Officials: Dana Graves, DDS, DMSc, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Temple University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania